CLINICAL TRIAL: NCT00136565
Title: A Phase II Study Evaluating the Efficacy and Safety of Bortezomib (Velcade™) Combined With ACVBP Regimen in Patients With Previously Untreated Peripheral T-cell Lymphoma
Brief Title: Study of Bortezomib Combined With ACVBP in Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Collaborators: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNH05-1T; Janssen: i061-341-03; Eudract: 2005-001563-66
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: peripheral T-cell lymphomas; bortezomib; ACVBP regimen
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Bortezomib; Doxorubicin; Prednisone; Cyclophosphamide; Vindesine; Bleomycin

ARMS (1):
- Experimental (Experimental): Velcade, Doxorubicine, Cyclophosphamide, Vindesine, Bleomycin, Prednisone
  Interventions: Drug: Velcade; Drug: Doxorubicin; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Vindesine; Drug: Bleomycin

INTERVENTIONS:
Drug: Velcade — 1.5 mg/m², D1, D5, 4 cycles
Drug: Doxorubicin — 75 mg/m², D1, 4 cycles
Drug: Prednisone — 60 mg/m², D1-D5, 4 cycles
Drug: Cyclophosphamide — 1200 mg/m², D1, 4 cycles
Drug: Vindesine — 2 mg/m², D1, D5, 4 cycles
Drug: Bleomycin — 10 mg, D1, D5, 4 cycles

SUMMARY:
The purpose of this study is to determine the efficacy and the safety profile and toxicity of a combination of Velcade™ (bortezomib) with a standard chemotherapy regimen (ACVBP [doxorubicin, cyclophosphamide, vindesine, bleomycin, and prednisone]) in the treatment of previously untreated patients with peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
This is a multicentric, open-label, non-randomized, non-competitive clinical study, evaluating the efficacy and safety of V-ACVBP chemotherapy in previously untreated patients aged from 18 to 65 years with peripheral T-lymphoma.

It is anticipated that 60 subjects will be enrolled over two years (from June 2005 to May 2007).

The duration of the treatment period is approximately 28 weeks and patients are followed until death.

The total duration of the study is expected to be 5 years (from June 2005 to May 2010).

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated non-cutaneous peripheral T-cell lymphoma, including human T-cell lymphotropic virus type 1 (HTLV-1) related T-cell lymphoma, and natural killer (NK)-cell lymphoma.
* Ages 18 to 65 years.
* Life expectancy > 3 months.
* Written informed consent.

Exclusion Criteria:

* B-cell lymphoma or other subtype of T-cell lymphoma including anaplastic large cell lymphoma AKL(+), lymphoblastic lymphoma and primary cutaneous T-cell lymphoma.
* Any previous therapy for lymphoma except for short-term corticosteroids before inclusion.
* Inability to tolerate the ACVBP regimen according to investigator's judgement.
* Positive serology for HIV.
* Poor renal function (creatinin > 150 µmol/l within 14 days before enrollment), poor liver function (total bilirubin > 30 µmol/l, transaminases > 2.5 upper normal limit [UNL] within 14 days before enrollment), unless these abnormalities are related to the lymphoma.
* Poor bone marrow reserve as defined by neutrophils < 1.5 G/l or platelets < 100 G/l within 14 days before enrollment, unless these abnormalities are related to the lymphoma.
* Patient with >= grade 2 peripheral neuropathy non-related to lymphoma.
* Any central nervous system (CNS) disease.
* CNS or meningeal involvement by the lymphoma.
* Any serious active disease or comorbidity according to the investigator's decision.
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumours or stage 0 (in situ) cervical carcinoma.
* Known hypersensitivity to bortezomib, boron or mannitol.
* Contraindication to any cytotoxic drug contained in chemotherapy regimen.
* Pregnant or lactating women or women of childbearing potential not willing to use an adequate method of birth control (i.e. hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of study.
* Men not agreeing to take adequate contraceptive precautions during the study.
* Treatment with investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Adult patient under tutelage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01-08 (Actual); Primary Completion 2011-04-18 (Actual); Study Completion 2011-04-18 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 2 years
  percentage of patients alive with no event, events being defined as disease progression, institution of a new treatment for the lymphoma, relapse after complete response (CR), or death from any cause

SECONDARY OUTCOMES:
Complete response rate unconfirmed (CR+CR uncertain) | 2 years
  percentage of patients with complete response
Partial response (PR) rate | 2 years
  percentage of patients with partial response
Progression free survival (PFS) | 2 years
  Duration of survival without progression
Duration of response in complete responders (CR + CRu) | 2 years
Overall survival (OS) | 2 years
  Percentage of patients alive
Number of SAE | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Coiffier, MD, Study Chair — Hospices Civils de Lyon, Lyon, France; Alain Delmer, MD, Principal Investigator — Centre Hospitalier Robert Debré
Locations (5):
- Groupe d'Etude des Lymphomes de l'Adulte, Yvoir, Belgium
- France (4):
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Goy A, Younes A, McLaughlin P, Pro B, Romaguera JE, Hagemeister F, Fayad L, Dang NH, Samaniego F, Wang M, Broglio K, Samuels B, Gilles F, Sarris AH, Hart S, Trehu E, Schenkein D, Cabanillas F, Rodriguez AM. Phase II study of proteasome inhibitor bortezomib in relapsed or refractory B-cell non-Hodgkin's lymphoma. J Clin Oncol. 2005 Feb 1;23(4):667-75. doi: 10.1200/JCO.2005.03.108. Epub 2004 Dec 21. PMID 15613697
- [Background] O'Connor OA, Wright J, Moskowitz C, Muzzy J, MacGregor-Cortelli B, Stubblefield M, Straus D, Portlock C, Hamlin P, Choi E, Dumetrescu O, Esseltine D, Trehu E, Adams J, Schenkein D, Zelenetz AD. Phase II clinical experience with the novel proteasome inhibitor bortezomib in patients with indolent non-Hodgkin's lymphoma and mantle cell lymphoma. J Clin Oncol. 2005 Feb 1;23(4):676-84. doi: 10.1200/JCO.2005.02.050. Epub 2004 Dec 21. PMID 15613699
- [Background] Orlowski RZ. Proteasome inhibitors in cancer therapy. Methods Mol Biol. 2005;301:339-50. doi: 10.1385/1-59259-895-1:339. PMID 15917644
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org